CLINICAL TRIAL: NCT01085799
Title: Effectiveness of a Post-deworming Education Intervention to Reduce Soil-transmitted Helminth Infections and Absenteeism in Grade 5 School-children in a Community of Extreme Poverty, Peruvian Amazon
Brief Title: Education Intervention to Reduce Helminth Infections and Absenteeism in Grade 5 School-children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Theresa W. Gyorkos, PhD, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEN-09-214; HOA-80064 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Infections
Keywords: Educational activities; Cluster-randomized controlled trial; Albendazole; Deworming; School-age children; Peru; Ascaris lumbricoides; Trichuris trichiura; Hookworm; STH infections; Intestinal helminth infections
MeSH Terms: conditions — Infections; Trichuriasis; Ancylostomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education Intervention (Experimental): Groups of schools receiving the health education intervention
  Interventions: Behavioral: Health Education Intervention
- Control Schools - Regular curriculum (No Intervention): Groups of schools not receiving the health education intervention

INTERVENTIONS:
Behavioral: Health Education Intervention — This is a health hygiene education strategy which encourages the pro-active role of both teachers and students and changes in attitudes and practices with the aim of keeping the level of parasite infection low, through increased knowledge.
  Arms: Health Education Intervention

SUMMARY:
To efficiently control soil-transmitted helminths (Ascaris, Trichuris, and hookworm), WHO, PAHO, and others recommend the inclusion of an education strategy in school-based deworming programs. However, the effectiveness of such a strategy on the rate of STH re-infection and on education indicators, such as absenteeism, remains to be fully understood. The proposed research aims to evaluate the effectiveness of a post-deworming education intervention targeted to Grade 5 school children enrolled in Belén's schools using a cluster-randomized trial design. Results will be used to inform school-based deworming programs in Peru and other similar endemic areas in Latin America and, indeed, around the world.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys enrolled in Grade 5 in eligible schools located in the Belén district of Iquitos, Peru. Eligible schools have a minimum of 10 boys and 10 girls enrolled in grade 5.
* Informed written consent obtained from the parents or legal guardian of the child.
* Verbal assent from child.

Exclusion Criteria:

* Parents (or guardians) refusing participation of their child.
* Child who refuses to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1101 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Soil-transmitted helminth re-infection (Ascaris, Trichuris, or Hookworm). | 4 months post-deworming

SECONDARY OUTCOMES:
Absenteeism rate. | During the first 4 months following deworming
Eggs per grams reduction rate. | 4 months post-deworming
Weight gain (kg) | 4 months post-deworming
Height gain (cm) | 4 months post-deworming

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W. Gyorkos, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Martín Casapía, MD, MPH, Study Director — Asociación Civil Selva Amazónica
Locations (1):
- Asociación Civil Selva Amazónica, Iquitos, Loreto, Peru